CLINICAL TRIAL: NCT01928199
Title: A Single Center, Randomized, Double-blind Controlled Trial of Sitagliptin Versus Placebo to Reduce the Incidence and Severity of New-onset Diabetes After Kidney Transplant
Brief Title: Efficacy Study of Sitagliptin to Prevent New-onset Diabetes After Kidney Transplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201306111; 50669 (Other Grant/Funding Number: Merck)
Record Dates: First submitted 2013-08-20; First posted 2013-08-23 (Estimated); Results first posted 2021-06-29 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Posttransplant Diabetes Mellitus
Keywords: diabetes; transplant; kidney
MeSH Terms: conditions — Diabetes Mellitus | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin (Active Comparator): Sitaglipitin tablets will be administered orally for 3 months from randomization
  Initial dose will be 100mg/daily, adjusted per renal function:
  Creatinine clearance > or = 50mL/min: 100mg/day Creatinine clearance > or = 30 and <50mL/min: 50mg/day Creatinine clearance <30 mL/min or on dialysis: 25mg/day
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): Placebo tablets (identical to active comparator in appearance) will be administered orally for 3 months. Starting dose and adjustment based on renal function will be identical to active comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether sitagliptin is effective in preventing the development of new-onset diabetes after kidney transplant (NODAT). Up to one-third of previously non-diabetic patients develop NODAT after a kidney transplant. Corticosteroids and calcineurin inhibitors are two commonly utilized anti-rejection medications that contribute to diabetes development through multiple mechanisms; including decreased insulin production by the pancreas. Sitagliptin is an oral medication that results in increased insulin secretion. We hypothesize that administration of sitagliptin to transplant recipients identified to be at risk for diabetes development will reduce the incidence and severity of NODAT.

DETAILED DESCRIPTION:
This will be a single-center, randomized, double-blind trial to evaluate the efficacy of sitagliptin to prevent the development of new-onset diabetes after transplant (NODAT) in previously non-diabetic patients with post-operative hyperglycemia following living-donor or deceased-donor kidney transplant. In this trial, previously non-diabetic adult patients with hyperglycemia (random blood sugar >200mg/dL) in the first 72 hours following kidney transplant will be screened to determine eligibility based on inclusion/exclusion criteria. Patients that meet study entry criteria will be stratified based on HbA1c (<5.7 or 5.7-6.4%) and randomized in a 1:1 ratio to one of two treatment groups: sitagliptin versus placebo. Fifty patients (25 per group) will be enrolled. Dosing period will be 3 months at which time study drug will be discontinued and patients will be followed for an additional 3 month period.

Study visits will occur at 0, 1, 3 and 6 months. A HbA1c and 2-hour oral glucose tolerance test (OGTT) will be obtained at the 3 and 6 month study visit.

Screening period (Visit 1)

All patients presenting for living-donor or deceased donor kidney transplant will have a medical history, medication history, vital signs, height, weight, body mass index, physical exam, random blood sugar (BS), HbA1c and EKG done as part of routine pre-transplant protocol at Barnes Jewish Hospital. Patients with hyperglycemia, defined as a random blood sugar ≥ 200 mg/dL, in the first 72 hours after kidney transplant will be screened to determine eligibility for the study based on inclusion and exclusion criteria.

Randomization (Visit 2)

Patients meeting study entry criteria and consenting to study participation will be stratified based on HbA1c (<5.7 or 5.7-6.4%) and block randomized in blocks of eight in a 1:1 ratio to sitagliptin versus placebo. Sitagliptin dose will be 100mg/day, adjusted per creatinine clearance and tolerability. Patients will be instructed by a licensed diabetic educator on proper measurement and recording of fasting and post-prandial blood sugars. Subjects will be provided a log, standard glucometer and testing strips to maintain a blood sugar log post-discharge. Visit 2 will occur within 24 hours after Visit 1.

Drug dosing period (Visits 3-4)

Sitagliptin or placebo will be continued until 3 months post-transplant, at which time study medication will be discontinued and collected from the subject. At the 1 and 3 month visits, vital signs, height, weight, and BMI will be obtained. A physical exam will be performed. Blood sugar logs provided by the patient will be reviewed and adverse effects recorded. At the 3 month visit (Visit 4), a HbA1c, 2-hour OGTT, fasting C-peptide and insulin level will be obtained.

Follow-up (Visit 5)

At the 6 month final visit, 3 months following discontinuation of study medication, vital signs, height, weight, BMI, HbA1c, 2-hour OGTT, fasting C-peptide and insulin level will be obtained. A physical exam will be performed. Blood sugar logs provided by the patient will be reviewed and adverse effects recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 yo) recipient of living-donor or deceased donor kidney transplant
2. Blood sugar ≥ 200 mg/dL in first 72 hours after transplant
3. No history of diabetes or prior treatment with insulin or oral hypoglycemic agents

Exclusion Criteria:

1. A1c of ≥6.5% measured immediately pre-transplant
2. Recipient of simultaneous kidney-pancreas, kidney-liver, kidney-heart, or kidney-lung transplant
3. Prior non-renal solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-09; Primary Completion 2020-06 (Actual); Study Completion 2020-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rowena Delos Santos, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Background] Yates CJ, Fourlanos S, Hjelmesaeth J, Colman PG, Cohney SJ. New-onset diabetes after kidney transplantation-changes and challenges. Am J Transplant. 2012 Apr;12(4):820-8. doi: 10.1111/j.1600-6143.2011.03855.x. Epub 2011 Nov 28. PMID 22123607
- [Background] Caillard S, Eprinchard L, Perrin P, Braun L, Heibel F, Moreau F, Kessler L, Moulin B. Incidence and risk factors of glucose metabolism disorders in kidney transplant recipients: role of systematic screening by oral glucose tolerance test. Transplantation. 2011 Apr 15;91(7):757-64. doi: 10.1097/TP.0b013e31820f0877. PMID 21336240
- [Background] Chakkera HA, Knowler WC, Devarapalli Y, Weil EJ, Heilman RL, Dueck A, Mulligan DC, Reddy KS, Moss AA, Mekeel KL, Mazur MJ, Hamawi K, Castro JC, Cook CB. Relationship between inpatient hyperglycemia and insulin treatment after kidney transplantation and future new onset diabetes mellitus. Clin J Am Soc Nephrol. 2010 Sep;5(9):1669-75. doi: 10.2215/CJN.09481209. Epub 2010 Jun 17. PMID 20558559
- [Background] Herman GA, Bergman A, Stevens C, Kotey P, Yi B, Zhao P, Dietrich B, Golor G, Schrodter A, Keymeulen B, Lasseter KC, Kipnes MS, Snyder K, Hilliard D, Tanen M, Cilissen C, De Smet M, de Lepeleire I, Van Dyck K, Wang AQ, Zeng W, Davies MJ, Tanaka W, Holst JJ, Deacon CF, Gottesdiener KM, Wagner JA. Effect of single oral doses of sitagliptin, a dipeptidyl peptidase-4 inhibitor, on incretin and plasma glucose levels after an oral glucose tolerance test in patients with type 2 diabetes. J Clin Endocrinol Metab. 2006 Nov;91(11):4612-9. doi: 10.1210/jc.2006-1009. Epub 2006 Aug 15. PMID 16912128
- [Background] Lane JT, Odegaard DE, Haire CE, Collier DS, Wrenshall LE, Stevens RB. Sitagliptin therapy in kidney transplant recipients with new-onset diabetes after transplantation. Transplantation. 2011 Nov 27;92(10):e56-7. doi: 10.1097/TP.0b013e3182347ea4. No abstract available. PMID 22067216

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin: Sitaglipitin tablets will be administered orally for 3 months from randomization
  Initial dose will be 100mg/daily, adjusted per renal function:
  Creatinine clearance > or = 50mL/min: 100mg/day Creatinine clearance > or = 30 and <50mL/min: 50mg/day Creatinine clearance <30 mL/min or on dialysis: 25mg/day
  Sitagliptin
- Placebo: Placebo tablets (identical to active comparator in appearance) will be administered orally for 3 months. Starting dose and adjustment based on renal function will be identical to active comparator
  Placebo
Period: Overall Study
Arm/Group | Sitagliptin | Placebo
Started | 32 | 29
Completed | 27 | 23
Not Completed | 5 | 6
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 3 | 5

BASELINE CHARACTERISTICS:
Population: We measured baseline hemoglobin A1c
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 32 | 29 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 24 | 50
  >=65 years | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.71 (12.63) | 51.81 (16.54) | 51.34 (13.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 17 | 17 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 22 | 23 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 29 | 61
Hemoglobin A1c [Mean (Standard Deviation); unit: percent] | 5.27 (0.46) | 5.13 (0.41) | 5.20 (0.44)

OUTCOME MEASURES:

1. Primary Outcome: 2-hour Oral Glucose Tolerance Test-derived Blood Sugar
Description: Change in 2-hour OGTT-derived blood sugar will be measured at three months and again at six months. These are 3 month OGTT results
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 27 | 23
mg/dL | 141.00 (62.44) | 165.22 (72.03)

2. Secondary Outcome: Normal 2-hour Oral Glucose Tolerance Test-derived Blood Sugar
Description: Number of subjects who have normal 2-hour oral glucose tolerance test-derived blood sugar will be measured at 3 months
Time Frame: 3 months
Population: Lower numbers for this due to drop out
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 27 | 23
Participants | 16 | 10

3. Secondary Outcome: 6 Month OGTT Result (Completion of Washout From Study Drug)
Description: We tested another OGTT at 6 months into study, after a 3 month washout from the study drug. Study drug was discontinued after the 3 month OGTT was completed.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 27 | 23
mg/dL | 174.38 (77.93) | 171.86 (83.69)

4. Other Pre Specified Outcome: Hemoglobin A1c, 3 Month
Description: Measurement of Hemoglobin A1c at 3 months of being on study drug/placebo
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 27 | 23
percentage of glycosylated hemoglobin | 5.52 (0.58) | 5.78 (0.85)

5. Other Pre Specified Outcome: Hemoglobin A1c, 6 Month
Description: This is the result of hemoglobin A1c measured 3 months after stopping study drug/placebo, tested at the 6 month study time point
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 27 | 23
percentage of glycosylated hemoglobin | 5.91 (0.84) | 5.79 (0.69)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events related to admissions described were part of post transplant events, determined not due to medication side effects
Arm/Group | Sitagliptin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/29
Serious Adverse Events (participants affected / at risk) | 3/32 | 3/29
Other Adverse Events (participants affected / at risk) | 0/32 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=32) | Placebo (N=29)
Urine leak (Renal and urinary disorders) | 1 (1) | 0 (0) — Patient experienced urine leak during study period, requiring admission and repair
Volume overload (Cardiac disorders) | 1 (1) | 0 (0) — Admission during study period for volume overload requiring diuresis
Right arm weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient was evaluated for right arm weakness; no other significant findings additionally
Hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1) — Patient underwent elective hernia repair during study period
shortness of breath (Cardiac disorders) | 0 (0) | 1 (1) — Patient was evaluated for shortness of breath during study period; no other additional events
Bilateral native nephrectomy (Renal and urinary disorders) | 0 (0) | 1 (1) — Patient underwent elective bilateral native nephrectomy surgery during study period

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT01928199/Prot_SAP_000.pdf